CLINICAL TRIAL: NCT04972175
Title: A Randomized Controlled Pilot Study to Assess the Pharmacokinetics, Pharmacodynamics, and Closed-loop Efficacy of BC LisPram Compared to Rapid Insulin in Pump-treated Adults With Type 1 Diabetes
Brief Title: Safety and Efficacy of BC LisPram
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Tsoukas (Network)
Collaborators: Adocia (Industry)
Responsible Party: Sponsor-Investigator, Michael Tsoukas, Principal Investigator, Applied Medical Informatics Research Inc.
Organization: Applied Medical Informatics Research Inc. (Network)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00050920; Pro00050920 (Other: Research Ethics Board - Advarra)
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rapid Insulin lispro - Conventional bolus (Active Comparator): Participants will use subcutaneously-delivered rapid insulin (lispro) through pump therapy.
  Interventions: Drug: 50-Hour Intervention - Rapid Insulin lispro
- BC LisPram - Conventional bolus (Experimental): Participants will use subcutaneously-delivered BC LisPram through pump therapy.
  Interventions: Drug: 50-Hour Intervention - BC LisPram
- BC LisPram - Dual wave bolus (Experimental): Participants will use subcutaneously-delivered BC LisPram through pump therapy. During dual wave bolusing, 50% of the prandial bolus is delivered immediately, and the other 50% delivered over the next 30 minutes.
  Interventions: Drug: 50-Hour Intervention - BC LisPram

INTERVENTIONS:
Drug: 50-Hour Intervention - Rapid Insulin lispro — Subcutaneous-delivery of insulin lispro using pump therapy.
  Arms: Rapid Insulin lispro - Conventional bolus
Drug: 50-Hour Intervention - BC LisPram — Subcutaneous-delivery of BC LisPram using pump therapy.
  Arms: BC LisPram - Conventional bolus; BC LisPram - Dual wave bolus

SUMMARY:
This pilot study is a 50-hour randomized, open-label, crossover study in an inpatient setting assessing the safety, pharmacodynamics, pharmacokinetics, and closed-loop efficacy of i) BC LisPram delivery and ii) rapid insulin delivery.

DETAILED DESCRIPTION:
Subjects will be randomized to intervention sequences. The first 6 participants will be randomly allocated to a sequence of three treatments composed of (i) treatment with active comparator insulin lispro, (ii) treatment with BC LisPram, and (iii) treatment with BC LisPram (dual wave bolus). The following 10 participants will be randomly allocated to a sequence of either two or three treatments. Each treatment period will last 50 hours. PK/PD assessment will be performed under an open-loop system and will be followed by a 24 hour of closed-loop assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age.
* Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Insulin pump therapy for at least 3 months, with daily insulin needs ranging between 30 and 80 U.
* Most recent HbA1c ≤ 9.5% (over the last two months).
* Effective birth control in female participants of childbearing potential. Medically acceptable contraception methods include condom, pills, and intrauterine device.

Exclusion Criteria:

* Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2, GLP-1, Metformin, Acarbose, etc....).
* Current use of glucocorticoid medication.
* Use of medication that alters gastrointestinal motility.
* Planned or ongoing pregnancy.
* Breastfeeding individuals
* Severe hypoglycemic episode within one month of admission.
* Severe diabetic ketoacidosis episode within one month of admission.
* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* Known hypersensitivity to any of the study drugs or their excipients.
* Allergy to paracetamol (acetaminophen).
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Clinically abnormal significant values for haemato, biochemistry, or urinalysis screening test as judged by the Principle Investigator for underlying disease.
* Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of Pramlintide | Breakfast, lunch, dinner from 0 to 4 hours
  Area under the pramlintide concentration-time curve
Pharmacokinetics of Insulin | Breakfast, lunch, dinner from 0 to 4 hours
  Area under the insulin concentration-time curve
Pharmacokinetics of Paracetamol | Breakfast and dinner from 0 to 4 hours
  Area under the paracetamol concentration-time curve
Glucose Pharmacodynamics | Breakfast, lunch and dinner from 0 to 4 hours
  Area under the sensor glucose concentration-time curve
Glucagon Pharmacodynamics | Breakfast and dinner from 0 to 4 hours
  Area under the plasma glucagon concentration-time curve
Hypoglycaemic episodes | 0 to 50 hours
  Number of hypoglycaemic episodes during the 0 to 50 hour period.
Gastrointestinal symptoms | 0 to 50 hours
  Frequency of gastrointestinal symptoms during the 0 to 50 hour period.
Local tolerability at pump injection site | 0 to 50 hours
  Local tolerability at pump injection site during the 0 to 50 hour period.
Incidence of adverse event | 0 to 50 hours
  Number of adverse events during the 0 to 50 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, MD, Principal Investigator — Applied Medical Informatics Research Inc.
Locations (1):
- Hygea Medical Clinic, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No